CLINICAL TRIAL: NCT00694941
Title: A Phase II Multi-centre, Extension Study to Investigate the Long Term Safety of ONO-2506PO in Patients Diagnosed With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-2506POE015
Record Dates: First submitted 2008-06-06; First posted 2008-06-11 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: ONO-2506PO; Amyotrophic Lateral Sclerosis; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- E (Experimental): ONO-2506PO in the presence of Riluzole
  Interventions: Drug: ONO-2506PO

INTERVENTIONS:
Drug: ONO-2506PO — 1200mg QD / 5 years

SUMMARY:
The objective of this study is to investigate the long term safety of ALS patients taking ONO-2506PO.

DETAILED DESCRIPTION:
This is an extension study which consists of two phases:

Double-blind phase; Patients will continue to take blinded study medication, as allocated in study ONO-2506POE014 by the central randomization system, in the presence of stable standard Riluzole therapy, until un-blinding of the study results.

Open label phase; Patients who were allocated to ONO-2506PO in the ONO-2506POE014 study will be offered entry into the open label phase of ONO-2506POE015 study and will continue to take 1200 mg of ONO-2506PO for the duration of their participation in the study, in the presence of stable standard Riluzole therapy. Patients who were allocated to placebo in ONO-2506POE014 study will be withdrawn from ONO-2506POE015 study, but will continue to be followed up by their site with standard care.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients with diagnosis of ALS over the age of 18 years.
* Previous randomization and completion of the last visits in ONO-2506POE014 study.
* Patients whom the investigator has no concern and judges tolerable for the continued treatment with ONO-2506PO and Riluzole from a risk and benefit point of view.

Exclusion Criteria:

* A clinically relevant medical history or presence of cardiovascular, gastrointestinal, renal, hepatic, endocrine/metabolic, neurologic, lymphatic, haematologic, immunologic, musculoskeletal, connective tissue, dermatologic, genito/urinary, psychiatric diseases or disorders that, in the opinion of the investigator may pose an unwarranted risk to the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Oct 2013
Death | Oct 2013
Tracheotomy or permanent assisted ventilation | Oct 2013

CONTACTS AND LOCATIONS:
Overall Officials: Tomohiro Kuwayama, Study Director — Ono Pharma UK
Locations (25):
- Belgium (2):
  - Prof. Maloteaux, UCL Saint-Luc, Brussels
  - Prof. Wim Robberecht, UZ Leuven, Leuven
- France (6):
  - Prof. Alain Destee, Hopital Roger Salengro - Clinique Neurologique, Neurologie A, Lille
  - Prof. Philippe Couratier, Hopital Duruytren, Limoges
  - Prof. Jan Pouget, Hopital de la Timone, Marseille
  - Prof. William Camu, Hopital de Chauliac, Montpellier
  - Prof. Claude Desnuelle, Hopital 1-Archet 1, Nice
  - Prof. Vincent Meininger, Hopital LaPitie Salpetriere, Paris
- Germany (8):
  - Dr. Thomas Meyer, Charite Campus Virchow, ALS Ambulanz, Berlin
  - Prof. Torsten Grehl, Neurologische Ambulanz Universitatsklinik Bergmannsheil, Bochum
  - Professor Dieter Heuss, Poliklinik der Universitat Erlangen-Nurnberg, Neurologische Klinik, Erlangen
  - Prof. Stephan Zierz, Martin Luther Universitat Halle-Wittenberg, Klinikum der Medizinischen Fakultat, Universitatsklinik und Poliklinik fur Neurologie, Halle
  - Prof. Reinhard Dengler, Medizinische Hochschule Hannover, Neurologische Klinik, Hanover
  - Prof Gian Domenico Borasio, Interdisziplinares Zentrum fur Palliativmedizin, München
  - Prof. Albert Ludolph, Klinik und Poliklinikfur Neurologie der Universitat Ulm-Univeritatsklinikum Ulm, Ulm
  - Dr. Berthold Schrank, Deutsche Klinik fur Diagnostik, Fachbereich Neurologie, Wiesbarden
- Italy (3):
  - Prof. Vincenzo Silani, Dipartimento di Neurologia e Laboratorio di Neuroscienze - Universita di Milano - IRCCS - Istituto Auxologico Italiano, Milan
  - Dr. Gabriele Mora, Divisione di Neuroriabilitazione II - Fondazione Salvatore Maugeri - IRCCS, Pavia
  - Prof. Adriano Chio, Dipartimento di Neuroscienze - Divisione di Neurologia II - Azienda Ospedaliera S. Giovanni Battista - Molinette, Torino
- Netherlands (2):
  - Prof Marianne de Visser, Academic Medical Centre (AMC) Amsterdam - Dept of Neurology, Amsterdam
  - Prof. Leonard H Van Den Berg, University Medical Center Utrecht, Utrecht
- Dr. Markus Weber, Kantonsspital St. Gallen, Muskelzentrum/ALS Clinic, Sankt Gallen, Switzerland
- United Kingdom (3):
  - Prof. Nigel Leigh, Academic Neuroscience Centre, London
  - Prof. Douglas Mitchell, Royal Preston Hospital, Preston
  - Dr. Chris McDermott, Royal Hallamshire Hospital, Sheffield